CLINICAL TRIAL: NCT05129540
Title: Foot Orthoses in Patients with Chronic Sciatica Caused by Lumbar Disc Herniation: a Randomized Clinical Trial
Brief Title: Foot Orthoses in Patients with Sciatica
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Large number of loss of participats.
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Pedro V. Munuera-Martínez, Full Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCIATICA AND FOOT
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2023-11

CONDITIONS: Chronic Sciatica; Foot Deformity
MeSH Terms: conditions — Foot Deformities | interventions — Foot Orthoses

STUDY DESIGN:
Intervention Model Description: Two groups of people with chronic sciatica caused by lumbar disc herniation will be included. Patients in group A will be given treatment with custom-made foot orthoses. Patients in group B will be given treatment with placebo orthoses.
Who Masked: Participant, Investigator
Masking Description: Custom-made foot orthoses and placebo orthoses will have similar appearance for participants. The investigator who record data by means of questionnaires will not know which group the patients belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Custom-made foot orthoses group (Experimental): Custom-made foot orthoses will be applied to participants in this arm. The orthoses will consist on a 3-mm thick polypropylene layer from heel to just proximal to the metatarsal heads, and a cover layer of polyethylene foam from heel to toe tips. Both materials will be adapted to the foot positive casts that will be obtained from all participants.
  Interventions: Device: Custom-made foot orthosis
- Placebo group (Placebo Comparator): The placebo orthoses will consist on a 3-mm thick polyethylene foam layer from heel to toe tips and a 0.8-mm thick resin layer from heel to just proximal to the metatarsal heads. None of the materials will be adapted to the foot positive casts.
  Interventions: Device: Placebo orthosis

INTERVENTIONS:
Device: Custom-made foot orthosis — The foot orthoses for group A will be custom made using phenolic foam molds of the feet. They consist of a polypropylene layer of 3 mm from heel to just proximal to the metatarsal heads, and an upper sheet of 30 Shore A polyethylene foam.
  Other Names: Foot orthotics; Insole
  Arms: Custom-made foot orthoses group
Device: Placebo orthosis — A flat insole made of the same material as the upper layer of the custom-made foot orthoses used for group "custom-made foot orthosis".
  Arms: Placebo group

SUMMARY:
Chronic sciatica is a frequent problem whose symptoms could be related to the abnormal stresses applied to the musculoskeletal system during the gait cycle due to foot alterations.

The objectives of this study are to describe the main foot alterations in patients with chronic sciatica, and to evaluate whether foot orthoses can help alleviate this pain. Patients with chronic sciatica caused by lumbar disc herniation will be recruited and randomly allocate to one of both groups: one group that will be treated with custom-made foot orthoses, and one group that will be treated with a placebo orthotic device. Quality of life, pain in low-back, lower limb and foot, and disability caused by foot pain will be recorded at baseline, and after a two-month follow-up period.

DETAILED DESCRIPTION:
A multi-centre randomised controlled clinical trial has been designed according to the CONSORT guidelines. The design was carried out by the research group (5 researchers, Ph.D and Degree in Podiatry, from the University of Seville and 2 researchers, Medicine Doctors, from the university hospital "Virgen de Valme", in Seville, Spain). The patients will be diagnosed and recruited from the aforementioned hospital. The data will be gathered in the Clinical Area of Podiatry of the University of Seville.

The main inclusion criteria will be to have a medical diagnosis of chronic sciatica (CS) caused by lumbar disc herniation (LDH). All participants who voluntarily take part in the study will be given an informative document where the nature, objectives, and potential risks of the investigation are explained. When the participants have read it and any doubts have been resolved, the informed consent will be given for them to sign.

Firstly, clinical and demographic data will be collected, including age, gender, weight, height, years since diagnosis and current pharmacological management. Patients with CS will be explored and the Foot Posture Index (FPI) (a validated method for quantifying standing foot posture), and the Manchester scale for hallux valgus will be recorded for both the right and left foot. Plantar pressure will be obtained using the footscan® Advanced Pressure Measurement System (RsScan Lab LTD, UK). Standard podiatric care will be provided to the patients at the assessment session and when finished the follow up three months later, if needed. Participants will be requested not to have further foot interventions.

After the biomechanical examination, phenolic foam molds will be made of the patient's feet under weight-bearing conditions. The patient's foot will be manipulated before being introduced into the phenolic foam so as to place the subtalar joint in the most neutral position possible, always maintaining the forefoot plantar plane parallel to the ground. In the case of FPI values between +6 and +12, the examiner will hold the distal third of the participant's leg and apply external rotational force to the leg until the mirror of the pedoscope shows incipient loss of the first ray footprint that is, that the first metatarsal begins to elevate. At that moment, the examiner will stop applying external rotational force to the leg. The examiner will repeat this manoeuvre several times, as the external rotation applied to the foot in contact with the glass will be the same as that applied when introducing the foot into the phenolic foam. The same procedure but with internal rotation of the leg will be carried out for FPI values between -12 to -1. For feet with FPI values between 0 and +5, the examiner's hands will apply resistance against pronation or supination in order to maintain the foot in a normal posture.

For foot orthoses delivery one researcher will verify the fitting of the orthosis to the patient's foot. Then the orthosis will be set into shoes. Finally, the participants will be asked if the insoles cause them pain or discomfort in every session. Both interventions have the same protocol.

The software AleatorMetod.xls, available at www4.ujaen.es/~mramos/EPIP/AleatorMetod.xls, will be used to randomly allocate the participants into two groups, and this allocation will be concealed in envelopes. The simple randomisation process will be carried out according to the order of appointment, so that the first patient treated will be number 1. The participants themselves will choose the day and time to attend the Podiatric Clinical Area without knowing the order number that participants have or the corresponding random assignment. Group A will be the experimental group and will receive the custom-made foot orthoses and Group B will be the control group and will be given the placebo treatment. Both groups will be followed up for 3 months, and the data related to foot pain, be recorded monthly by phone. This phone call will remind the participants to appropriately use the orthoses during the follow-up period.

The primary outcome is pain within the foot, lower extremity and lumbar region. Visual analogue scale will be used to record pain at baseline and at the end of the follow-up period, and self-reported pain intensity once a month by phone call will be assessed with an 11-point NPRS with 0 = no pain to 10 = pain as bad as it can be.

Secondary outcomes will be disability related to foot pain, and quality of life. Disability related to foot pain will be measured using the Manchester Foot Pain and Disability Index (MFPDI) at baseline and at the end of the follow-up period. The values of this index range from 0 to 38, with higher values corresponding to greater disability. The SF-12 questionnaire will be used to collect data about the quality of life. This has values between 0 and 100, with higher values corresponding to a lower quality of life.

All the participants will be blinded, as will not know what group belong to and the type of orthoses that will be given in the study (intervention or placebo). Patients will only be informed that the research will evaluate this treatment to manage pain in patients with CS caused by LDH. The participants will be requested to use the foot orthoses assigned seven days a week for a minimum of eight hours per day for three months. The researcher who performs the measurements at days 0, 30, 60, and 90 will not be the same researcher who conducts the randomisation, adapts the foot orthoses, and gives them to the participants. Thus, researchers will be blinded as well. Adverse events will be recorded as part of the monitoring and appropriate safety measures. The participants will be asked about any problems with the foot orthoses and their adaptation to the footwear.

The minimum sample size was calculated using the following formula to compare mean values between populations:

n = (2s^2 (z_(α/2) + z_β))/d^2, where s2 is the sample variance, α is the type I error, β is the type II error, and d is the minimum difference to be detected. According to previous studies, the variance of the visual analogue scale for pain is equal to 400, and the difference found is 16. Therefore, the following result was obtained: n = (2s^2 (z_(α/2) + z_β))/d^2 = 〖2 ∙ 400 ∙ (1.96+0.84)〗^2/16^2 = 24.5 = 25 Thus, at least 25 people will be needed in each group to compare the mean values. In this study, 100 patients will be initially recruited, with 50 in each group, in consideration of possible losses.

The analysis of the data will becarried out using the statistical software IBM SPSS Statistics (IBM, Armonk, NY, USA). The descriptive data will provide the mean values and the standard deviations or the absolute frequencies and percentages depending on whether the variables are scalar or categorical. Shapiro-Wilk tests will be conducted for the inferential analysis to determine the most appropriate test to use. When the data show a normal distribution by groups, a t-test for independent samples will be carried out. Mann-Whitney's U test will be used for the independent samples when there is no normal distribution. For those study variables that will be measured four times, the tests will be conducted in pairs for related samples as well. The t-test will be used if the variables show a normal distribution in the four measurements, and Wilcoxon's signed-rank test will be used for related samples when do not. When statistically significant differences are found according to the P-value, the effect size will be calculated using Cohen's d or Rosenthal's r to analyse the magnitude of the differences. The differences will be classified according to the following for both parameters: below 0.2: no effect; 0.2-0.5: small effect; 0.5-0.8: medium effect; and above 0.8: large effect. The analyses will be based on an intention-to-treat data set.

In the case of the variables for which randomisation produces differences between groups at the initial assessment, repeated-measures analyses of covariance (ANCOVAs) with the baseline scores as covariates will be performed to enable comparisons of post-intervention data after adjusting for those differences in the initial scores.

The confidence level a priori is 95%. For missing data (participant withdrawal or interim missing data), the convenience of several missing data models (i.e., 'missing at random', 'missing completely at random' or 'missing not at random') will be classified by the trial personnel (according to available trial data). The most appropriate missing data model will be selected.

Data monitoring will be evaluated in collaboration with an external Statistician, who will also review all the issues related to data collection and analysis during the research process.

ELIGIBILITY:
Inclusion Criteria:

* Having lumbar and/or lower extremity pain.
* Having a medical diagnosis of chronic sciatica caused by lumbar disc herniation.

Exclusion Criteria:

* Ulcers within the foot.
* Diabetes mellitus.
* Pregnancy.
* Cognitive deterioration.
* Previous osteoarticular foot surgery.
* Concomitant inflammatory rheumatic disease.
* Need for walking assistance.
* Being treated with foot orthotics.
* Refuse to use appropriated and health footwear (with no more than a 3 cm drop, wide and spacious with removable, laced or velcro insole, posterior buttress, medial-lateral stability, and flexibility in metatarsophalangeal area to allow dorsiflexion).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Rate of Lumbar pain | 3 months
  Rate of pain perceived in the lumbar region. Visual analogue scale will be used to record pain at baseline and at the end of the follow-up period, and self-reported pain intensity once a month by phone call will be assessed with an 11-point NPRS with 0 = no pain to 10 = pain as bad as it can be.
Rate of ower limb pain | 3 months
  Rate of pain perceived in the posterior surface of the lower extremity. Visual analogue scale will be used to record pain at baseline and at the end of the follow-up period, and self-reported pain intensity once a month by phone call will be assessed with an 11-point NPRS with 0 = no pain to 10 = pain as bad as it can be.
Rate of foot pain | 3 months
  Rate of pain perceived in the foot and ankle region. Visual analogue scale will be used to record pain at baseline and at the end of the follow-up period, and self-reported pain intensity once a month by phone call will be assessed with an 11-point NPRS with 0 = no pain to 10 = pain as bad as it can be.

SECONDARY OUTCOMES:
Rate of Quality of life | 3 months
  Self-perceived quality of life assessed by the Short Form 12 Health Survey (SF-12). This has values between 0 and 100, with higher values corresponding to a lower quality of life.
Rate of disability related to the foot | 3 months
  Disability related to foot pain will be measured using the Manchester Foot Pain and Disability Index (MFPDI) at baseline and at the end of the follow-up period. The values of this index range from 0 to 38, with higher values corresponding to greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro V Munuera-Martínez, Ph.D, Principal Investigator — University of Seville
Locations (1):
- Department of Podiatry, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blunt SB, Richards PG, Khalil N. Foot dystonia and lumbar canal stenosis. Mov Disord. 1996 Nov;11(6):723-5. doi: 10.1002/mds.870110620. PMID 8914101
- [Background] Dananberg HJ, Guiliano M. Chronic low-back pain and its response to custom-made foot orthoses. J Am Podiatr Med Assoc. 1999 Mar;89(3):109-17. doi: 10.7547/87507315-89-3-109. PMID 10095332
- [Background] Bird AR, Bendrups AP, Payne CB. The effect of foot wedging on electromyographic activity in the erector spinae and gluteus medius muscles during walking. Gait Posture. 2003 Oct;18(2):81-91. doi: 10.1016/s0966-6362(02)00199-6. PMID 14654211
- [Background] Al Kutobi ZTA, Al Omari WRS. The effect of chronic sciatica on the knee and ankle joints. Qatar Medical Journal. 2003; 12(2): 98-100
- [Background] Shabat S, Gefen T, Nyska M, Folman Y, Gepstein R. The effect of insoles on the incidence and severity of low back pain among workers whose job involves long-distance walking. Eur Spine J. 2005 Aug;14(6):546-50. doi: 10.1007/s00586-004-0824-z. Epub 2005 Jan 25. PMID 15668775
- [Background] Pomares Avalos AJ, Lopez Fernandez R, Zaldivar Perez DF. [Validation of the Oswestry disability scale for low back pain in patients with chronic back pain. Cienfuegos, 2017-2018]. Rehabilitacion (Madr). 2020 Jan-Mar;54(1):25-30. doi: 10.1016/j.rh.2019.10.003. Epub 2019 Dec 24. Spanish. PMID 32007179
- [Background] Eslami M, Tanaka C, Hinse S, Farahpour N, Allard P. Eslami, M. Effect of foot wedge positions on lower-limb joints, pelvis and trunk angle variability during single-limb stance. Foot (Edinburg) 2006; 16(4): 208-213.
- [Background] Khamis S, Yizhar Z. Effect of feet hyperpronation on pelvic alignment in a standing position. Gait Posture. 2007 Jan;25(1):127-34. doi: 10.1016/j.gaitpost.2006.02.005. Epub 2006 Apr 18. PMID 16621569
- [Background] Parker N, Greenhalgh A, Chockalingam N, Dangerfield PH. Positional relationship between leg rotation and lumbar spine during quiet standing. Stud Health Technol Inform. 2008;140:231-9. PMID 18810029
- [Background] Pinto RZ, Souza TR, Trede RG, Kirkwood RN, Figueiredo EM, Fonseca ST. Bilateral and unilateral increases in calcaneal eversion affect pelvic alignment in standing position. Man Ther. 2008 Dec;13(6):513-9. doi: 10.1016/j.math.2007.06.004. Epub 2007 Oct 1. PMID 17910932
- [Background] Ghahreman A, Ferch RD, Rao P, Chandran N, Shadbolt B. Recovery of ankle dorsiflexion weakness following lumbar decompressive surgery. J Clin Neurosci. 2009 Aug;16(8):1024-7. doi: 10.1016/j.jocn.2008.10.017. Epub 2009 May 9. PMID 19428255
- [Background] van Tulder M, Peul W, Koes B. Sciatica: what the rheumatologist needs to know. Nat Rev Rheumatol. 2010 Mar;6(3):139-45. doi: 10.1038/nrrheum.2010.3. Epub 2010 Feb 9. PMID 20142811
- [Background] Cambron JA, Duarte M, Dexheimer J, Solecki T. Shoe orthotics for the treatment of chronic low back pain: a randomized controlled pilot study. J Manipulative Physiol Ther. 2011 May;34(4):254-60. doi: 10.1016/j.jmpt.2011.04.004. Epub 2011 May 5. PMID 21621727
- [Background] Tateuchi H, Wada O, Ichihashi N. Effects of calcaneal eversion on three-dimensional kinematics of the hip, pelvis and thorax in unilateral weight bearing. Hum Mov Sci. 2011 Jun;30(3):566-73. doi: 10.1016/j.humov.2010.11.011. Epub 2011 Apr 2. PMID 21459469
- [Background] O'Leary CB, Cahill CR, Robinson AW, Barnes MJ, Hong J. A systematic review: the effects of podiatrical deviations on nonspecific chronic low back pain. J Back Musculoskelet Rehabil. 2013;26(2):117-23. doi: 10.3233/BMR-130367. PMID 23640312
- [Background] Farokhmanesh K, Shirzadian T, Mahboubi M, Shahri MN. Effect of foot hyperpronation on lumbar lordosis and thoracic kyphosis in standing position using 3-dimensional ultrasound-based motion analysis system. Glob J Health Sci. 2014 Jun 17;6(5):254-60. doi: 10.5539/gjhs.v6n5p254. PMID 25169004
- [Background] Resende RA, Deluzio KJ, Kirkwood RN, Hassan EA, Fonseca ST. Increased unilateral foot pronation affects lower limbs and pelvic biomechanics during walking. Gait Posture. 2015 Feb;41(2):395-401. doi: 10.1016/j.gaitpost.2014.10.025. Epub 2014 Nov 3. PMID 25468683
- [Background] Park K. Effects of wearing functional foot orthotic on pelvic angle among college students in their 20s with flatfoot. J Phys Ther Sci. 2017 Mar;29(3):438-441. doi: 10.1589/jpts.29.438. Epub 2017 Mar 22. PMID 28356626
- [Background] Castro-Mendez A, Munuera PV, Albornoz-Cabello M. The short-term effect of custom-made foot orthoses in subjects with excessive foot pronation and lower back pain: a randomized, double-blinded, clinical trial. Prosthet Orthot Int. 2013 Oct;37(5):384-90. doi: 10.1177/0309364612471370. Epub 2013 Jan 17. PMID 23327838
- [Background] Yazdani F, Razeghi M, Karimi MT, Salimi Bani M, Bahreinizad H. Foot hyperpronation alters lumbopelvic muscle function during the stance phase of gait. Gait Posture. 2019 Oct;74:102-107. doi: 10.1016/j.gaitpost.2019.08.022. Epub 2019 Aug 31. PMID 31499403
- [Background] Kuo FC, Cai DC, Liau BY. Foot Arch Support Effect on Lumbo-Pelvic Kinematics and Centre of Pressure Excursion During Stand-to-Sit Transfer in Different Foot Types. Journal of Medical and Biological Engineering. 2020; 40:169-178
- [Background] Marchesini N, Ricci UM, Soda C, Teli M. Acute bilateral foot drop due to lumbar disc herniation treated by bilateral interlaminar approach: case report and literature review. Br J Neurosurg. 2023 Aug;37(4):899-901. doi: 10.1080/02688697.2020.1713992. Epub 2020 Jan 20. PMID 31955631
- [Background] Ali HM. Relationship between Lumbar Herniated Disc with Flat Feet. Sys Rev Pharm 2020;11(11):1804-1806.
- [Background] Chou MC, Huang JY, Hung YM, Perng WT, Chang R, Wei JC. Flat foot and spinal degeneration: Evidence from nationwide population-based cohort study. J Formos Med Assoc. 2021 Oct;120(10):1897-1906. doi: 10.1016/j.jfma.2020.12.019. Epub 2021 Jan 7. PMID 33423898
- [Background] Hornestam JF, Arantes PMM, Souza TR, Resende RA, Aquino CF, Fonseca ST, da Silva PLP. Foot pronation affects pelvic motion during the loading response phase of gait. Braz J Phys Ther. 2021 Nov-Dec;25(6):727-734. doi: 10.1016/j.bjpt.2021.04.005. Epub 2021 May 4. PMID 34020879
- [Background] Kararti C, Bilgin S, Dadali Y, Buyukturan B, Buyukturan O, Bek N. Are Biomechanical Features of the Foot and Ankle Related to Lumbopelvic Motor Control? J Am Podiatr Med Assoc. 2021 May 1;111(3):Article_13. doi: 10.7547/18-065. PMID 31625760
- [Background] Tanaka J, Takamori Y, Shiokawa T, Shibata R, Nobutou S, Shirachi H, Yamamoto T. Drop foot due to lumbar degenerative disease: Painless drop foot is difficult to recover. Clin Neurol Neurosurg. 2021 Jul;206:106696. doi: 10.1016/j.clineuro.2021.106696. Epub 2021 May 23. PMID 34059400